CLINICAL TRIAL: NCT06048302
Title: A Phase 1, Open-label, Single-dose, Parallel-group Study to Evaluate the Plasma Pharmacokinetics and Safety of Obicetrapib in Participants With Moderate Hepatic Impairment Relative to Participants With Normal Hepatic Function
Brief Title: PK and Safety in Participants Taking Obicetrapib With Moderate Hepatic Impairment Relative to Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Collaborators: Veranex (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TA-8995-12
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, single-dose, parallel-group study to evaluate the plasma PK and safety of obicetrapib in participants with moderate hepatic impairment relative to participants with normal hepatic function. The purpose of the study is to investigate the effect of moderate hepatic impairment on obicetrapib PK and safety in otherwise healthy participants after a single oral 10 mg dose of obicetrapib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparitor: Subjects with Moderate Hepatic Impairment (Active Comparator): 8 patients with hepatic impairment of moderate Child Pugh Category
  Interventions: Drug: Obicetrapib
- Active Comparator: Healthy Subjects (Other): Healthy volunteers will be matched with impaired hepatic function patients
  Interventions: Drug: Obicetrapib

INTERVENTIONS:
Drug: Obicetrapib — 1 single dose of obicetrapib
  Other Names: 10 mg tablet

SUMMARY:
To investigate the safety and pharmacokinetics in patients with moderate hepatic impairment compared to healthy participants after a single oral dose of obicetrapib (10 mg).

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single-dose, parallel-group study to evaluate the plasma PK and safety of obicetrapib in participants with moderate hepatic impairment relative to participants with normal hepatic function. The purpose of the study is to investigate the effect of moderate hepatic impairment on obicetrapib PK and safety in otherwise healthy participants after a single oral 10 mg dose of obicetrapib.

ELIGIBILITY:
Inclusion Criteria:

* A male or a female of non-childbearing potential.
* Women of childbearing potential (WOCBP) must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at the Screening Visit.
* Body mass index (BMI) of 17.5 to 42 kg/m2; with a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Cohort 1: Meet the criteria for Class B (moderate hepatic impairment) of the modified CPC. A diagnosis of hepatic dysfunction due to hepatocellular disease (and not secondary to any acute ongoing hepatocellular process) documented by medical history, physical examination (PE), liver biopsy, hepatic ultrasound, computerized tomography scan, or magnetic resonance imaging.
* Cohort 2: Will only enroll healthy volunteers with no hepatic impairment. "Healthy" is defined as no clinically relevant abnormalities identified by a detailed medical history, complete PE (including blood pressure [BP] and pulse rate measurement), 12-lead ECG or clinical laboratory tests performed during Screening.

Exclusion Criteria:

* Any condition possibly affecting drug absorption (e.g., gastrectomy). Uncomplicated cholecystectomy is allowed.
* History of or current positive results for human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV) or hepatitis C virus (HCV), including hepatitis B surface antigen (HbsAg) or hepatitis C Virus antibody (HCVAb).
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the Investigator's judgment, make the participant inappropriate for participation in the study.
* Participants with an estimated glomerular filtration rate (eGFR) value of ≤30 mL/min/1.73 m2, based on the 2021 Chronic Kidney Disease Epidemiology Collaboration equation during Screening. A single repeat assessment is permitted to assess eligibility, if needed.
* Previous administration of drugs or supplements known to be strong inducers or inhibitors of CYP3A4 within 7 days of planned dosing of obicetrapib on Day 1.
* Concurrent use of drugs or supplements that are known substrates of CYP3A that have narrow therapeutic indices (e.g., alfentanil, cyclosporine, dihydroergotamine, ergotamine, fentanyl including transdermal patch, pimozide, quinidine, sirolimus, tacrolimus) within 12 days prior to planned dosing of obicetrapib on Day 1.
* Participants on oral contraceptives and hormonal based contraceptives including implantable, intrauterine, intravaginal, transdermal or injectable form.
* Previous administration of an investigational drug within 30 days (or as determined by the local requirement) or within 5 half-lives of that investigational drug, prior to planned dosing of obicetrapib on Day 1.
* Known hypersensitivity to obicetrapib or its excipients.
* A positive urine drug test. Participants with moderate hepatic impairment (Cohort 1) will be eligible to participate if their urine drug test is positive with a drug for a prescribed condition that is not expected to interfere with the PK of obicetrapib. Positive urine drug tests for tetrahydrocannabinol (THC) will be allowed as long as the volunteer agrees to abstain from ingesting any THC-containing products for the duration of the study (including Out patient visits up to Day 28).
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to planned dosing of obicetrapib on Day 1.
* History of sensitivity to heparin or a history of heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the criteria in the Lifestyle considerations listed in the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Area under the curve from dosing time to infinity (AUC (0-inf)) for obicetrapib | 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168
  Blood samples collected
Area under curve from dosing time to last measurement (AUC (0-t)) for obicetrapib | 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168
  Blood Sample Collected
Observed maximum plasma concentration (Cmax) for Obicetrapib | 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 120, 168
  Blood Sample Collected

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nucleus Network, Saint Paul, Minnesota
  - The American Research Corporation, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No